CLINICAL TRIAL: NCT05654805
Title: Nutraceutical Improvement of Glucose Metabolism, NAFLD and Insulin Resistance by Oat-fiber Supplementation in Type 2 Diabetes Mellitus Patients
Acronym: NIMROD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Wilhelm-Doerenkamp-Foundation (Funding) (Unknown)
Responsible Party: Principal Investigator, Stefan Kabisch, Study physician, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIMROD
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes; NAFLD
Keywords: insoluble cereal fiber; insulin resistance; glucose tolerance; inflammation; incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Insulin Resistance; Inflammation

STUDY DESIGN:
Intervention Model Description: parallel-designed triple-blinded randomised placebo-controlled intervention study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: blinding applies to participants, study personnel and statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementation with insoluble cereal fiber (Active Comparator): Drinking powder supplement providing 7,5 grams of insoluble fiber per sachet, taken twice daily over a period of 12 weeks without any changes in dietary behavior, caloric intake or physical activity
  Interventions: Dietary Supplement: Drinking powder supplement
- Supplementation with placebo (Placebo Comparator): Drinking powder supplement providing no insoluble fiber, but maltodextrin, taken twice daily over a period of 12 weeks without any changes in dietary behavior, caloric intake or physical activity
  Interventions: Dietary Supplement: Drinking powder supplement

INTERVENTIONS:
Dietary Supplement: Drinking powder supplement — Drinking powder supplement, to be taken twice daily over 12 weeks

SUMMARY:
Cohort studies show an association between increased intake of insoluble (cereal) fiber and decreased risk for cardiovascular disease, type 2 diabetes (T2DM), non-alcoholic fatty liver disease (NAFLD), cancer, infectious and inflammatory disorders. Intervention studies, specifically addressing non-fermentable carbohydrates instead of their food sources (whole grain, pulses, legumes) are still sparse. Whole grain trials reported beneficial effects, but cannot pinpoint these benefits on fiber, as minerals, vitamins, grain protein and food matrix contribute to the metabolic results.

The antidiabetic effectiveness of cereal fiber might be explained by a) an increased secretion of incretins and other glucose-induced gastrointestinal hormones, b) an alteration of the gut microbiome, or c) a fermentation to short-chain fatty acids. Fermentable fibers (most of which are soluble) show these mechanisms, but lack strong diabetes-protective associations in cohort studies. In recent supplementation trials, insoluble, mostly non-fermentable fibers improved insulin resistance, glycemia and inflammation in patients with metabolic syndrome or prediabetes.

Between 2022-2024, we want to assess the effectiveness of insoluble, poorly fermentable cereal fiber in a shorter Intervention period in patients with high responsiveness (insulin-naïve overt type 2 diabetes mellitus with insulin resistance and NAFLD), using a fiber drinking supplement. Our triple-blinded RCT compares the metabolic effects and mechanistic outcomes of isocaloric treatments with 15 grams of oat-fiber supplement per day (vs. placebo) in 92 patients, covering an intervention period of 12 weeks.

DETAILED DESCRIPTION:
Cohort studies show an association between increased intake of insoluble (cereal) fiber and decreased risk for cardiovascular disease, type 2 diabetes (T2DM), non-alcoholic fatty liver disease (NAFLD), cancer, infectious and inflammatory disorders. Intervention studies, specifically addressing non-fermentable carbohydrates instead of their food sources (whole grain, pulses, legumes) are still sparse. Whole grain trials reported beneficial effects, but cannot pinpoint these benefits on fiber, as minerals, vitamins, grain protein and food matrix contribute to the metabolic results.

The antidiabetic effectiveness of cereal fiber might be explained by a) an increased secretion of incretins and other glucose-induced gastrointestinal hormones, b) an alteration of the gut microbiome, or c) a fermentation to short-chain fatty acids. Fermentable fibers (most of which are soluble) show these mechanisms, but lack strong diabetes-protective associations in cohort studies. In recent supplementation trials, insoluble, mostly non-fermentable fibers improved insulin resistance, glycemia and inflammation in patients with metabolic syndrome or prediabetes.

Between 2022-2024, we want to assess the effectiveness of insoluble, poorly fermentable cereal fiber in a shorter Intervention period in patients with high responsiveness (insulin-naïve overt type 2 diabetes mellitus with insulin resistance and NAFLD), using an oat fiber drinking supplement. Our triple-blinded RCT compares the metabolic effects and mechanistic outcomes of isocaloric treatments with 15 grams of oat-fiber supplement per day (vs. placebo) in 92 patients, covering an intervention period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* HOMA-IR > 2.5
* NAFLD (MR-S > 5,56 %)

Exclusion Criteria:

* insulin treatment
* diabetes type 1, 3 or 4
* severe cardiopulmonary, renal, inflammatory, gastrointestinal, psychiatric or endocrine disorder
* alcohol abuse or excess alcohol intake
* recent CVD event (< 3months)
* relevant liver disease other than NAFLD
* current cancer diagnosis or treatment
* allergy or incompatibility to the supplement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
change in liver fat content (MRS) | 12 weeks
  change in liver fat content (MRS)
change in glucose tolerance (mixed-meal test) | 12 weeks
  change in glucose tolerance (mixed-meal test)
change in insulin resistance (Matsuda) | 12 weeks
  change in insulin resistance (Matsuda)

SECONDARY OUTCOMES:
change in fasting glucose | 12 weeks
  change in fasting glucose
change in HbA1c | 12 weeks
  change in HbA1c
change in inflammation parameters (CRP, leucocytes, IL-6, IL-1ß, IL-18, IL-10, IL-22 | 12 weeks
  change in inflammation parameters (CRP, leucocytes, IL-6, IL-1ß, IL-18, IL-10, IL-22
change in incretins (GLP-1, GIP, PYY) | 12 weeks
  change in incretins (GLP-1, GIP, PYY)
change in FGF21 | 12 weeks
  change in FGF21
change in IGF-1 and its binding proteins | 12 weeks
  change in IGF-1 and its binding proteins

OTHER OUTCOMES:
change in secondary GI peptide hormons (GLP-2, PP, ghrelin, CCK) | 12 weeks
  change in secondary GI peptide hormons (GLP-2, PP, ghrelin, CCK)
change in fasting serum amino acid pattern | 12 weeks
  change in fasting serum amino acid pattern
change in faecal excretion of BCAA metabolites | 12 weeks
  change in faecal excretion of BCAA metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kabisch, Dr. med., Principal Investigator — Study physician
Locations (1):
- Charite University Hospital Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No